CLINICAL TRIAL: NCT05581407
Title: A Randomized First-in-human, Observer-blind, 3-arm Study to Evaluate Safety, Tolerability, and Immunogenicity of a Single Administration of TETRALITE, a Novel Adjuvanted, Low-dose Influenza Vaccine
Brief Title: Safety, Tolerability, and Immunogenicity of TETRALITE, a Novel Adjuvanted, Low-dose Influenza Vaccin
Acronym: TETRALITE-I
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LiteVax BV (Industry)
Collaborators: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2022-500681-98-00
Record Dates: First submitted 2022-09-27; First posted 2022-10-14 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2022-10

CONDITIONS: Influenza
Keywords: seasonal influenza vaccine; adjuvant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Comparison of licensed influenza vaccine with study vaccines combining 1/5 of the dose of the standard vaccine added with two different doses of LiteVax Adjuvant.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Licensed seasonal influenza vaccine (Active Comparator)
  Interventions: Biological: TETRALITE
- 1/5th of licensed seasonal influenza vaccine plus 1 mg LiteVax Adjuvant (Experimental)
  Interventions: Biological: TETRALITE
- 1/5th of licensed seasonal influenza vaccine plus 4 mg LiteVax Adjuvant (Experimental)
  Interventions: Biological: TETRALITE

INTERVENTIONS:
Biological: TETRALITE — LiteVax Adjuvanted Seasonal Influenza Vaccine

SUMMARY:
There is an obvious need for an affordable and more effective seasonal influenza vaccine. TETRALITE is a novel, inactivated, adjuvanted influenza vaccine combining a low dose of a licensed vaccine with the novel, potent LiteVax Adjuvant.

A licensed vaccine (Cohort 1) with a normal dose [15 ug per strain] and no adjuvant will be compared with two TETRALITE study vaccines with 1/5th of the licensed vaccine added with a low (Cohort 2) or high (Cohort 3) dose of LiteVax Adjuvant.

ELIGIBILITY:
Inclusion Criteria:

* Written signed informed consent obtained before any study-related activities.
* Aged 18 to 50 years inclusive, at the time of signing the ICF.
* Participants who are considered to be in good general health as determined by medical evaluation including medical history, physical examination and laboratory tests within 21 days prior to enrollment.
* Participants with a BMI within the range 18.5 to 35 kg/m2 inclusive at screening.
* Women who are not pregnant or breastfeeding (WOCBP).
* WOCBP must have a negative serum pregnancy test at screening and a negative urine pregnancy test before vaccination at Day 1.
* Participants who are willing and able to comply with the study procedures and are in the view of the investigator capable of completing the study.

Exclusion Criteria:

* History of previous laboratory confirmed influenza infection in the past 12 months, excluding laboratory confirmed COVID-19 infections, prior to the day of study vaccination.
* Positive (in the past, suspected or ongoing) for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, and human immunodeficiency virus (HIV) antibody.
* Past or current history of immune mediated and/or autoimmune diseases as indicated by the investigator, e.g. diabetes mellitus (type I or II, with the exception of gestational diabetes) and thyroid disease.
* Serious reactions to vaccines that preclude receipt of study vaccinations as determined by the investigator.
* Clinical conditions representing a contraindication for IM administration, as judged by the investigator, e.g. history of bleeding disorder (e.g. factor deficiency, coagulopathy, or platelet disorder requiring special precautions) or significant bruising or bleeding difficulties with IM administration or blood draws.
* History of confirmed hypersensitivity, allergy and/or anaphylaxis to eggs (ovalbumin or chicken proteins), squalene-based adjuvants, or other components of the study vaccine (neomycin, formaldehyde or octoxinol-9).
* Current history of uncontrolled medical illness (unstable for the past 3 months) as indicated by investigator, e.g. hypertension.
* Past or current history of any neurological disorder, e.g. Guillain-Barré syndrome and seizure disorder other than: 1) febrile seizures, 2) seizures secondary to alcohol withdrawal more than 3 years ago, or 3) seizures that have not required treatment within the last 3 years.
* History of asplenia, functional asplenia or any condition resulting in the absence or removal of the spleen.
* Active malignancy or malignancy within the past 5 years.
* Asthma that is unstable or required emergent care, urgent care, hospitalization or intubation during the past two years or that is expected to require the use of oral or intravenous corticosteroids.
* History of hereditary angioedema (HAE), acquired angioedema (AAE) or idiopathic forms of angioedema.
* History of idiopathic urticaria within the past year.
* History of heavy smoking, drug - or alcohol abuse/addiction (including alcohol dependence), or psychiatric condition (e.g. past or present psychoses; disorder requiring lithium; or within 5 years prior to administration of study vaccine, a history of suicide plan or attempt), which in investigator's opinion could compromise the participant's safety and/or compliance with the protocol.
* A rash, dermatological condition or tattoos that would, in the opinion of the investigator, interfere with injection local reaction rating.
* Prior seasonal or pandemic influenza vaccination in the 6 months before administration of study vaccine or planning to receive the influenza vaccination during the study period.
* Prior receipt of investigational pandemic influenza vaccine in the 3 months before administration of study vaccine or planning to receive such product during the study period.
* Prior receipt of a live attenuated vaccine in the 28 days prior to administration of study vaccine, or within 14 days for subunit or inactivated vaccines other than seasonal or pandemic influenza vaccination, excluding COVID-19 vaccine.
* Prior receipt of COVID-19 vaccine in the 7 days before administration of study vaccine, or planning to receive a COVID-19 vaccine during the first 14 days following study vaccination.
* Planning to receive a vaccine during the first 28 days following the administration of study vaccine, other than COVID-19 vaccine.
* Currently participating in another clinical study, or planning to participate in another study during the study period, or administration of any investigational drug or medical device in the 4 weeks prior to study vaccination.
* Prior receipt of blood, blood-derived products or immunoglobulins in the 6 months prior to administration of study vaccine, or planning to receipt such product during the study period.
* Use of drugs that can affect immune response such as systemic corticosteroids (excluding topical preparations and inhaled preparations) or immunosuppressive drugs in the 30 days before study vaccination and/or in the first 28 days following study vaccination, with the exceptions that a short course of corticosteroids ≤10 days duration, or a single injection for a self-limited condition at least 2 weeks prior to enrolment will not exclude study participation.
* Current intake of drugs that increase bleeding risk, e.g. anticoagulant medication (coumarin derivatives, low molecular weight heparin, DOAC).
* Current anti-tuberculosis prophylaxis or therapy.
* Use of non-steroidal anti-inflammatory drugs (NSAIDs) and/or planning a medical procedure under full anesthesia on the day of study vaccination and/or in the first 14 days following study vaccination with the exception of a medical indication.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-08-03 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single, intramuscular injection with TETRALITE | 6 months
  Monitoring of systemic adverse reactions
Safety and tolerability of a single, intramuscular injection with TETRALITE | 6 months
  Monitoring of local adverse reactions

SECONDARY OUTCOMES:
Immunogenicity of a single, intramuscular injection with TETRALITE | 9 months
  Monitoring haemagglutination inhibition (HI) antibody titres against the 4 influenza strains
Immunogenicity of a single, intramuscular injection with TETRALITE | 9 months
  Monitoring virus neutralisation (VN) antibody titres against the 4 influenza strains

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Leroux-Roels, PhD, Principal Investigator — CEVAC, University Hospital Ghent, Belgium
Locations (1):
- CEVAC, University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided